CLINICAL TRIAL: NCT00326014
Title: A Study of the Glaukos Trabecular Micro-Bypass Stent in Combination With Cataract Surgery in Open Angle Glaucoma Subjects.
Brief Title: A Study of the Trabecular Micro-Bypass Stent in Combination With Cataract Surgery in Open Angle Glaucoma Subjects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-002
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Open-Angle Glaucoma
Keywords: Open angle; Glaucoma; Cataract; Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Device: iStent

INTERVENTIONS:
Device: iStent — Glaucoma Surgery
  Other Names: Glaukos iStent

SUMMARY:
To evaluate the safety and efficacy of a new trabecular bypass that is implanted in conjunction with cataract surgery in open angle glaucoma subjects.

DETAILED DESCRIPTION:
Glaukos Corporation conducted a clinical research study at multiple investigational sites within Europe (8)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subject on at least one glaucoma medication
* Patient requiring cataract surgery and an intraocular lens implantation

Exclusion Criteria:

* Prior glaucoma procedures (eg trabeculectomy, viscocanalostomy, ALT, SLT, shunt implant, collagen implant, cyclo destructive procedures etc)
* Angle closure glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-04; Primary Completion 2008-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Head of clinical Affairs, Study Director — Glaukos Corporation
Locations (8):
- Germany (5):
  - Klinik Vincentinum, Augsburg
  - Universitats Augenklinik, Freiburg im Breisgau
  - Rotkreuz Krankenhaus, München
  - Klinikum Neubrandenburg, Neubrandenburg
  - Augenaerztliche Gemeinschaftspraxis, Weinheim
- Spain (2):
  - Clinico San Carlos, Madrid
  - Instituto Oftalmológico de Aragón, Zaragoza
- Augenklinik Kantonsspital, Winterthur, Switzerland

REFERENCES:
- [Background] Spiegel D, Wetzel W, Neuhann T, Stuermer J, Hoeh H, Garcia-Feijoo J, Martinez-De-La-Casa JM, Garcia-Sanchez J. Coexistent primary open-angle glaucoma and cataract: interim analysis of a trabecular micro-bypass stent and concurrent cataract surgery. Eur J Ophthalmol. 2009 May-Jun;19(3):393-9. doi: 10.1177/112067210901900311. PMID 19396784
- [Background] Spiegel D, Garcia-Feijoo J, Garcia-Sanchez J, Lamielle H. Coexistent primary open-angle glaucoma and cataract: preliminary analysis of treatment by cataract surgery and the iStent trabecular micro-bypass stent. Adv Ther. 2008 May;25(5):453-64. doi: 10.1007/s12325-008-0062-6. PMID 18594784